CLINICAL TRIAL: NCT00596713
Title: Epidemiology of Sleep Disturbances Among the Adult Population of the Sao Paulo City
Status: Completed | Type: Observational
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Prof. Dr. Lia Azeredo-Bittencourt, Prof. Dr., Associação Fundo de Incentivo à Pesquisa
Other Study IDs: 0593/06
Record Dates: First submitted 2008-01-09; First posted 2008-01-17 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: general population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Both genders aged 20 to 80 years and living in private households in the city of São Paulo. Pregnant or lactating women, people with physical or mental impairment and workers in night shifts are not part of the population of interest.

SUMMARY:
Sleep disturbances are of great relevance within the context of public health as they affect a sizable portion of the population with far reaching consequences. Many automobile and labor accidents as well as poor school and work performance can be traced to sleep disturbances, which are also linked to cardiovascular disease, metabolic syndrome, and psycho-cognitive alterations.

OBJECTIVES:

1. Establish the epidemiologic profile of sleep disturbances among the adult population of the city of Sao Paulo in 2007;
2. Investigate associations between sleep patterns and disturbances in that population, taking into account the following variables: social-demographic status, anthropometrics, clinical, activity/rest cycle, eating and physical activity habits, mood disturbances, sexual dysfunction in males, alcoholism, drug addiction, genetic markers, biochemical, hematological, endocrine, immunologic and inflammatory indicators;
3. assess the compatibility of the results collected in the current study with those of epidemiologic sleep investigations of said city carried out in 1987 and 1995 with the aim of determining the secular sleep disturbance trend.

METHODS:

The two-stage cluster randomized sample included 1100 individuals of the city of Sao Paulo, representing the population proportionally to gender, age groups and social classes. Data were amassed as follows:

1. the application of home and institution questionnaires;
2. description of the sleep patterns and disturbances through polysomnography and actigraphy, performed at the Sleep Institute;
3. collection of peripheral blood for biochemical, hematologic, endocrine and genetic assays.

STATISTICS:

Subsequent to double typing (inputting) and analysis of data consistency, descriptive and analytical statistical assessments will be performed with the aim of describing patterns of sleep disturbances associated to the explanatory variables under investigation. In the light of bi-varied analysis, predictive/explanatory multivaried models were adjusted.

ELIGIBILITY:
Inclusion Criteria:

* Both genders aged 20 to 80 years and living in private households in the city of São Paulo.

Exclusion Criteria:

* Pregnant or lactating women
* People with physical or mental impairment: and
* Workers in night shifts.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population of Sao Paulo city
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
sleep disorders | 1 night

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio S Silva, PhD, Principal Investigator — Associacao Fundo de Incentivo a Psicofarmcologia
Locations (1):
- AFIP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Maluly M, Dal Fabbro C, Andersen ML, Herrero Babiloni A, Lavigne GJ, Tufik S. Sleep bruxism and its associations with insomnia and OSA in the general population of Sao Paulo. Sleep Med. 2020 Nov;75:141-148. doi: 10.1016/j.sleep.2020.06.016. Epub 2020 Jun 20. PMID 32858352
- [Derived] Dokkedal-Silva V, Oliveira MGM, Galduroz JCF, Tufik S, Andersen ML. The effect of sleep medications on prospective and retrospective memory: a population-based study. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Jan 10;104:110043. doi: 10.1016/j.pnpbp.2020.110043. Epub 2020 Jul 16. PMID 32682875
- [Derived] Nunes RA, Mazzotti DR, Hirotsu C, Andersen ML, Tufik S, Bittencourt L. The association between caffeine consumption and objective sleep variables is dependent on ADORA2A c.1083T>C genotypes. Sleep Med. 2017 Feb;30:210-215. doi: 10.1016/j.sleep.2016.06.038. Epub 2016 Nov 15. PMID 28215251
- [Derived] Roizenblatt S, Souza AL, Palombini L, Godoy LM, Tufik S, Bittencourt LR. Musculoskeletal Pain as a Marker of Health Quality. Findings from the Epidemiological Sleep Study among the Adult Population of Sao Paulo City. PLoS One. 2015 Nov 24;10(11):e0142726. doi: 10.1371/journal.pone.0142726. eCollection 2015. PMID 26600201
- [Derived] de Godoy LB, Palombini LO, Martinho Haddad FL, Rapoport DM, de Aguiar Vidigal T, Klichouvicz PC, Tufik S, Togeiro SM. New insights on the pathophysiology of inspiratory flow limitation during sleep. Lung. 2015 Jun;193(3):387-92. doi: 10.1007/s00408-015-9714-x. Epub 2015 Apr 1. PMID 25827757
- [Derived] Castro LS, Poyares D, Leger D, Bittencourt L, Tufik S. Objective prevalence of insomnia in the Sao Paulo, Brazil epidemiologic sleep study. Ann Neurol. 2013 Oct;74(4):537-46. doi: 10.1002/ana.23945. Epub 2013 Sep 16. PMID 23720241
- [Derived] Maluly M, Andersen ML, Dal-Fabbro C, Garbuio S, Bittencourt L, de Siqueira JT, Tufik S. Polysomnographic study of the prevalence of sleep bruxism in a population sample. J Dent Res. 2013 Jul;92(7 Suppl):97S-103S. doi: 10.1177/0022034513484328. Epub 2013 May 20. PMID 23690359
- [Derived] Manzotte T, Guindalini C, Mazzotti DR, Palombini L, de Souza AL, Poyares D, Bittencourt LR, Tufik S. The human leucocyte antigen DQB1*0602 allele is associated with electroencephelograph differences in individuals with obstructive sleep apnoea syndrome. J Sleep Res. 2013 Apr;22(2):217-22. doi: 10.1111/jsr.12005. Epub 2012 Nov 9. PMID 23136848
- [Derived] Mazzotti DR, Guindalini C, Pellegrino R, Barrueco KF, Santos-Silva R, Bittencourt LR, Tufik S. Effects of the adenosine deaminase polymorphism and caffeine intake on sleep parameters in a large population sample. Sleep. 2011 Mar 1;34(3):399-402. doi: 10.1093/sleep/34.3.399. PMID 21359089
- [Derived] Santos-Silva R, Bittencourt LR, Pires ML, de Mello MT, Taddei JA, Benedito-Silva AA, Pompeia C, Tufik S. Increasing trends of sleep complaints in the city of Sao Paulo, Brazil. Sleep Med. 2010 Jun;11(6):520-4. doi: 10.1016/j.sleep.2009.12.011. Epub 2010 May 21. PMID 20494615
- [Derived] Guindalini C, Colugnati FA, Pellegrino R, Santos-Silva R, Bittencourt LR, Tufik S. Influence of genetic ancestry on the risk of obstructive sleep apnoea syndrome. Eur Respir J. 2010 Oct;36(4):834-41. doi: 10.1183/09031936.00146809. Epub 2010 Mar 11. PMID 20223916